CLINICAL TRIAL: NCT03971422
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating Efficacy and Safety of Rozanolixizumab in Adult Patients With Generalized Myasthenia Gravis
Brief Title: A Study to Test Efficacy and Safety of Rozanolixizumab in Adult Patients With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG0003; 2019-000968-18 (EudraCT Number)
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Generalized Myasthenia Gravis
Keywords: UCB7665; generalized myasthenia gravis; rozanolixizumab; gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dosage Regimen 1 (Experimental): Study participants randomized to dosage regimen 1 will receive assigned dosage of rozanolixizumab at pre-specified time points during Treatment Period.
  Interventions: Drug: Rozanolixizumab
- Dosage Regimen 2 (Experimental): Study participants randomized to dosage regimen 2 will receive assigned dosage of rozanolixizumab at pre-specified time points during Treatment Period.
  Interventions: Drug: Rozanolixizumab
- Placebo (Placebo Comparator): Study participants randomized to this arm will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rozanolixizumab — Rozanolixizumab will be administered by subcutaneous infusion in dosage regimen 1 or 2.
  Other Names: UCB7665
  Arms: Dosage Regimen 1; Dosage Regimen 2
Other: Placebo — Subjects will receive placebo at pre-specified time points.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of the MycarinGstudy is to demonstrate the clinical efficacy and to assess safety and tolerability of rozanolixizumab in patients with generalized myasthenia gravis (MG).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥18 years of age, at the time of signing the informed consent
* Study participant has documented diagnosis of generalized myasthenia gravis (gMG) at Visit 1, based on study participant's history and supported by previous evaluations
* Study participant has a confirmed positive record of autoantibodies against acetylcholine receptor (AChR) or muscle-specific kinase (MuSK) at Screening (Visit 1).The presence of autoantibodies may be confirmed with repeat testing at Visit 1
* Study participant has Myasthenia Gravis Foundation of America (MGFA) Class II to IVa at Visit 1
* Study participant with a Myasthenia Gravis-Activities of Daily Living (MG-ADL) score of at least 3 (with ≥3 points from non-ocular symptom) AND a quantitative myasthenia gravis (QMG) score of at least 11 at Visit 1 and at Baseline (Visit 2)
* Study participant is considered for additional treatment such as intravenous immunoglobulin g (IVIg) or plasma exchange (PEX) by the Investigator

Exclusion Criteria:

* Study participant has a known history of hyperprolinemia
* Study participant has a clinically relevant active infection (eg, sepsis, pneumonia, or abscess) in the opinion of the Investigator, or had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to the first dose of investigational medicinal product (IMP)
* Study participant with a known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent tuberculosis infection (LTBI), or current/history of nontuberculous mycobacterial infection (NTMBI) will be excluded
* Study participant has experienced hypersensitivity reaction after exposure to other anti-neonatal Fc receptor (FcRn) drugs
* Study participant with severe (defined as Grade 3 on the Myasthenia Gravis-Activities of Daily Living (MG-ADL) scale) weakness affecting oropharyngeal or respiratory muscles, or who has myasthenic crisis or impending crisis at Visit 1 or Visit 2
* Study participant has a history of a solid organ transplant or hematopoietic stem cell/marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (112):
- United States (30):
  - Mg0003 50081, Phoenix, Arizona
  - Mg0003 50082, Scottsdale, Arizona
  - Mg0003 50072, Los Angeles, California
  - Mg0003 50092, Orange, California
  - Mg0003 50097, San Francisco, California
  - Mg0003 50099, San Francisco, California
  - Mg0003 50101, Aurora, Colorado
  - Mg0003 50088, Washington D.C., District of Columbia
  - Mg0003 50122, Miami, Florida
  - Mg0003 50120, Miami, Florida
  - Mg0003 50073, Tampa, Florida
  - Mg0003 50075, Augusta, Georgia
  - Mg0003 50323, Honolulu, Hawaii
  - Mg0003 50109, Chicago, Illinois
  - Mg0003 50114, Indianapolis, Indiana
  - Mg0003 50074, Fairway, Kansas
  - Mg0003 50121, Lexington, Kentucky
  - Mg0003 50110, Ann Arbor, Michigan
  - Mg0003 50102, Detroit, Michigan
  - Mg0003 50104, Rochester, Minnesota
  - Mg0003 50105, St Louis, Missouri
  - Mg0003 50077, New York, New York
  - Mg0003 50117, Charlotte, North Carolina
  - Mg0003 50086, Charlotte, North Carolina
  - Mg0003 50090, Winston-Salem, North Carolina
  - Mg0003 50076, Columbus, Ohio
  - Mg0003 50096, Philadelphia, Pennsylvania
  - Mg0003 50089, Philadelphia, Pennsylvania
  - Mg0003 50084, Charleston, South Carolina
  - Mg0003 50113, Houston, Texas
- Mg0003 40121, Brussels, Belgium
- Canada (4):
  - Mg0003 50067, Calgary
  - Mg0003 50066, Montreal
  - Mg0003 50070, Québec
  - Mg0003 50069, Toronto
- Czechia (2):
  - Mg0003 40125, Ostrava
  - Mg0003 40124, Prague
- Denmark (4):
  - Mg0003 40128, Aalborg
  - Mg0003 40127, Aarhus N
  - Mg0003 40126, Copenhagen
  - Mg0003 40489, Odense
- France (11):
  - Mg0003 40129, Bordeaux
  - Mg0003 40070, Clermont-Ferrand
  - Mg0003 40512, Garches
  - Mg0003 40510, Le Kremlin-Bicêtre
  - Mg0003 40360, Limoges
  - Mg0003 40426, Lyon
  - Mg0003 40130, Marseille
  - Mg0003 40017, Nantes
  - Mg0003 40132, Nice
  - Mg0003 40133, Paris
  - Mg0003 40131, Strasbourg
- Georgia (4):
  - Mg0003 20160, Tbilisi
  - Mg0003 20161, Tbilisi
  - Mg0003 20163, Tbilisi
  - Mg0003 20165, Tbilisi
- Germany (6):
  - Mg0003 40134, Essen
  - Mg0003 40140, Göttingen
  - Mg0003 40135, Gummersbach
  - Mg0003 40139, Jena
  - Mg0003 40078, Leipzig
  - Mg0003 40177, Münster
- Hungary (2):
  - Mg0003 40082, Kistarcsa
  - Mg0003 40178, Nyíregyháza
- Italy (7):
  - Mg0003 40283, Bologna
  - Mg0003 40149, Lazio
  - Mg0003 40144, Milan
  - Mg0003 40307, Napoli
  - Mg0003 40146, Pavia
  - Mg0003 40148, Roma
  - Mg0003 40150, Roma
- Japan (12):
  - Mg0003 20035, Bunkyō City
  - Mg0003 20068, Chiba
  - Mg0003 20078, Hanamaki-Shi
  - Mg0003 20079, Hiroshima
  - Mg0003 20075, Kobe
  - Mg0003 20071, Nagasaki
  - Mg0003 20074, Ōsaka-sayama
  - Mg0003 20067, Sapporo
  - Mg0003 20077, Sendai
  - Mg0003 20070, Shinjuku-Ku
  - Mg0003 20076, Shinjuku-Ku
  - Mg0003 20032, Suita
- Poland (4):
  - Mg0003 40155, Gdansk
  - Mg0003 40154, Lodz
  - Mg0003 40151, Lublin
  - Mg0003 40153, Poznan
- Russia (8):
  - Mg0003 20168, Krasnoyarsk
  - Mg0003 20027, Moscow
  - Mg0003 20169, Novosibirsk
  - Mg0003 20001, Saint Petersburg
  - Mg0003 20028, Saint Petersburg
  - Mg0003 20029, Saint Petersburg
  - Mg0003 20055, Saint Petersburg
  - Mg0003 20197, Samara
- Serbia (2):
  - Mg0003 40468, Belgrade
  - Mg0003 40467, Niš
- Spain (9):
  - Mg0003 40159, Barcelona
  - Mg0003 40160, Barcelona
  - Mg0003 40267, Barcelona
  - Mg0003 40157, L'Hospitalet de Llobregat
  - Mg0003 40161, Madrid
  - Mg0003 40162, Madrid
  - Mg0003 40341, Málaga
  - Mg0003 40350, Murcia
  - Mg0003 40308, San Sebastián de los Reyes
- Taiwan (4):
  - Mg0003 20080, Taichung
  - Mg0003 20081, Taipei
  - Mg0003 20086, Taipei
  - Mg0003 20082, Taoyuan District
- United Kingdom (2):
  - Mg0003 40175, London
  - Mg0003 40168, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Result] Bril V, Druzdz A, Grosskreutz J, Habib AA, Mantegazza R, Sacconi S, Utsugisawa K, Vissing J, Vu T, Boehnlein M, Bozorg A, Gayfieva M, Greve B, Woltering F, Kaminski HJ; MG0003 study team. Safety and efficacy of rozanolixizumab in patients with generalised myasthenia gravis (MycarinG): a randomised, double-blind, placebo-controlled, adaptive phase 3 study. Lancet Neurol. 2023 May;22(5):383-394. doi: 10.1016/S1474-4422(23)00077-7. PMID 37059507
- [Result] Habib AA, Sacconi S, Antonini G, Cortes-Vicente E, Grosskreutz J, Mahuwala ZK, Mantegazza R, Pascuzzi RM, Utsugisawa K, Vissing J, Vu T, Wiendl H, Boehnlein M, Greve B, Woltering F, Bril V. Efficacy and safety of rozanolixizumab in patients with muscle-specific tyrosine kinase autoantibody-positive generalised myasthenia gravis: a subgroup analysis of the randomised, double-blind, placebo-controlled, adaptive phase III MycarinG study. Ther Adv Neurol Disord. 2024 Sep 12;17:17562864241273036. doi: 10.1177/17562864241273036. eCollection 2024. PMID 39297052
- [Result] Kaminski HJ, Antozzi C, Habib AA, Pascuzzi RM, Sacconi S, Utsugisawa K, Vissing J, Regnault A, Hareendran A, Grimson F, Tarancon T, Bril V; MycarinG study investigators. Improvement in Patient-Reported Symptoms of Generalised Myasthenia Gravis With Rozanolixizumab in the Randomised Phase 3 MycarinG Study Using the MG Symptoms PRO. Eur J Neurol. 2025 Aug;32(8):e70231. doi: 10.1111/ene.70231. PMID 40755069
- [Result] Barnett-Tapia C, Cortes Vicente E, Pascuzzi RM, Utsugisawa K, Bloemers J, Grimson F, Tarancon T, Bril V; MycarinG study investigators. Measuring the effect of rozanolixizumab using the Myasthenia Gravis Impairment Index: analyses from the randomized phase 3 MycarinG study. J Neurol. 2025 Nov 8;272(12):752. doi: 10.1007/s00415-025-13480-8. PMID 41205003
- [Derived] Regnault A, Habib AA, Creel K, Kaminski HJ, Morel T. Clinical meaningfulness and psychometric robustness of the MG Symptoms PRO scales in clinical trials in adults with myasthenia gravis. Front Neurol. 2024 Jun 24;15:1368525. doi: 10.3389/fneur.2024.1368525. eCollection 2024. PMID 38978809
- [Derived] Matic A, Alfaidi N, Bril V. An evaluation of rozanolixizumab-noli for the treatment of anti-AChR and anti-MuSK antibody-positive generalized myasthenia gravis. Expert Opin Biol Ther. 2023 Jul-Dec;23(12):1163-1171. doi: 10.1080/14712598.2023.2296126. Epub 2023 Dec 28. PMID 38099334
- [Derived] Bril V, Benatar M, Andersen H, Vissing J, Brock M, Greve B, Kiessling P, Woltering F, Griffin L, Van den Bergh P; MG0002 Investigators. Efficacy and Safety of Rozanolixizumab in Moderate to Severe Generalized Myasthenia Gravis: A Phase 2 Randomized Control Trial. Neurology. 2021 Feb 9;96(6):e853-e865. doi: 10.1212/WNL.0000000000011108. Epub 2020 Nov 20. PMID 33219142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in Jun 2019 and concluded in Oct 2021.
Pre-assignment Details: Participant Flow refers to the Randomized Set. Two participants randomized to RLZ ~7mg/kg, were administered RLZ ~10mg/kg at baseline visit. So, these two participants were included in RLZ ~7 mg/kg group in randomized set, but in RLZ ~10 mg/kg group in safety set.
Groups:
- Placebo: Participants received placebo subcutaneously on a weekly basis over a 6-week Treatment Period. After 6-week Treatment Period, participants were followed for up to 8 weeks (up to Week 14).
- Rozanolixizumab ~7 mg/kg: Participants received rozanolixizumab (RLZ) equivalent to approximately 7 milligrams/kilogram (mg/kg), subcutaneously on a weekly basis over a 6-week Treatment Period. After 6-week Treatment Period, participants were followed for up to 8 weeks (up to Week 14).
- Rozanolixizumab ~10 mg/kg: Participants received rozanolixizumab equivalent to approximately 10 mg/kg, subcutaneously on a weekly basis over a 6-week Treatment Period. After 6-week Treatment Period, participants were followed for up to 8 weeks (up to Week 14).
Period: Overall Study
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Started | 67 | 66 | 67
Completed | 42 | 43 | 43
Not Completed | 25 | 23 | 24
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Lack of Efficacy | 5 | 1 | 1
Not completed — Adverse event, not fatal | 2 | 2 | 5
Not completed — Worsening of MG Symptoms | 1 | 4 | 2
Not completed — Roll over to MG0007 (NCT04650854) | 10 | 6 | 9
Not completed — Roll over to MG0004 (NCT04124965) | 7 | 8 | 6
Not completed — Due to COVID-19 pandemic | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Randomized Set (RS) which consisted of all study participants who were randomized and analyzed according to the treatment assigned instead of the actual treatment received.
Groups:
- Rozanolixizumab ~7 mg/kg: Participants received rozanolixizumab equivalent to approximately 7 mg/kg, subcutaneously on a weekly basis over a 6-week Treatment Period. After 6-week Treatment Period, participants were followed for up to 8 weeks (up to Week 14).
- Total: Total of all reporting groups
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg | Total
Number analyzed (Participants) | 67 | 66 | 67 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 50 | 49 | 51 | 150
  >=65 years | 16 | 17 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (17.7) | 53.2 (14.7) | 51.9 (16.5) | 51.8 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 39 | 35 | 121
  Male | 20 | 27 | 32 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 9 | 7 | 21
  Black | 1 | 0 | 4 | 5
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  White | 46 | 41 | 49 | 136
  Missing | 14 | 16 | 7 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 3 | 13
  Not Hispanic or Latino | 48 | 47 | 58 | 153
  Missing | 14 | 14 | 6 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 43 in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Score
Description: The Myasthenia Gravis Activities of Daily Living (MG-ADL) is an 8-item patient-reported outcome (PRO) instrument developed on the basis of the Quantitative Myasthenia Gravis (QMG). The MG-ADL targeted symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The total MG-ADL score was obtained by summing the responses to each individual item (8 items; Grades: 0, 1, 2, 3), where 0 represents no symptoms or impaired performance and 3 represents the most severe symptoms or impaired performance. The total score ranges from 0 to 24, with a higher score indicating more disability. A positive change in the score indicates worsening and a negative change indicates improvement.
Time Frame: Baseline and Day 43
Population: The Randomized Set consisted of all study participants who were randomized and analyzed according to the treatment assigned instead of the actual treatment received.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 66 | 67
units on a scale | -0.784 (0.488) | -3.370 (0.486) | -3.403 (0.494)
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab ~7 mg/kg; The parallel gatekeeping testing procedure with a truncated Hochberg test was used to control the familywise type I error rate at a 2-sided alpha level of 0.05; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — Confidence intervals and p-values are based on stage-wise inverse normal combination using the Lehmacher and Wassmer method; LS Mean Difference = -2.586, 95% CI 2-sided [-4.091 to -1.249] — Mixed model repeated measure (MMRM) ANCOVA model included treatment group, Baseline score, region, stratification factor (MuSK+ or AChR+) and treatment group by day (interaction term) as fixed factors and participant as a random effect
Statistical Analysis 2: Comparison: Placebo vs Rozanolixizumab ~10 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -2.619, 95% CI 2-sided [-3.994 to -1.163] — MMRM analysis of covariance (ANCOVA) model included treatment group, Baseline score, region, stratification factor (MuSK+ or AChR+) and treatment group by day (interaction term) as fixed factors and participant as a random effect

2. Secondary Outcome: Percentage of Participants Achieving Myasthenia Gravis-Activities of Daily Living (MG-ADL) Response at Day 43
Description: The MG-ADL is an 8-item PRO instrument developed on the basis of the QMG. The MG-ADL targeted symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The total MG-ADL score was obtained by summing the responses to each individual item (8 items; Grades: 0, 1, 2, 3), where 0 represents no symptoms or impaired performance and 3 represents the most severe symptoms or impaired performance. The total score ranges from 0 to 24, with a higher score indicating more disability. A positive change in the score indicates worsening and a negative change indicates improvement. Study participants were classified as responders at Day 43 if the value was at least a 2-point improvement (decrease) from Baseline at Day 43.
Time Frame: Day 43
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 66 | 67
percentage of participants | 28.4 | 68.2 | 61.2
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab ~7 mg/kg; Test type: Superiority; p < 0.001, Wald test — p-value is nominal. Confidence intervals and p-values are based on stage-wise inverse normal combination using the Lehmacher and Wassmer method; Odds Ratio (OR) = 5.765, 95% CI 2-sided [2.100 to 14.882] — The OR of responder rates is estimated and tested between treatment groups using logistic regression model with treatment group, Baseline MG-ADL score and stratification factor (MuSK+ or AChR+). An OR > 1 favours rozanolixizumab
Statistical Analysis 2: Comparison: Placebo vs Rozanolixizumab ~10 mg/kg; Test type: Superiority; p < 0.001, Wald test — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.273, 95% CI 2-sided [1.653 to 11.791] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline to Day 43 in Myasthenia Gravis-Composite (MG-C) Total Score
Description: MG-C scale is a validated assessment and scale tests 10 items with individual item being weighted differently. The items included ptosis/upward gaze (range: 0 [>45 second] - 3 [Immediate]), double vision on lateral gaze (range: 0 [>45 second] - 4 [Immediate]), eye closure (range: 0 [Normal] - 2 [severe weakness]), talking (range: 0 [Normal] - 6 [difficult to understand speech]), chewing (range: 0 [Normal] - 6 [gastric tube]), swallowing (range: 0 [Normal] - 6 [gastric tube]), breathing (range: 0 [Normal] - 9 [ventilator dependence]), neck flexion (range: 0 [Normal] - 4 [severe weakness]), shoulder abduction (range: 0 [Normal] - 5 [severe weakness]) and hip flexion (range: 0 [Normal] - 5 [severe weakness]), lower scores= lower disease activity. Total MG-C score was obtained by summing responses to each individual item and score ranges from 0 to 50, with lower scores indicating lower disease activity. A positive change indicates worsening and a negative change indicates improvement.
Time Frame: Baseline and Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 66 | 67
units on a scale | -2.029 (0.917) | -5.930 (0.916) | -7.554 (0.934)
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab ~7 mg/kg; A sequential testing procedure was used. The parallel gatekeeping testing procedure with a truncated Hochberg test was used to control the familywise type I error rate at a 2-sided alpha level of 0.05; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -3.901, 95% CI 2-sided [-6.634 to -1.245] — MMRM ANCOVA model included treatment group, Baseline score, region, stratification factor (MuSK+ or AChR+) and treatment group by day (interaction term) as fixed factors and participant as a random effect
Statistical Analysis 2: Comparison: Placebo vs Rozanolixizumab ~10 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -5.525, 95% CI 2-sided [-8.303 to -2.968] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline to Day 43 in Quantitative Myasthenia Gravis (QMG) Total Score
Description: The QMG is a validated assessment and the scale tested 13 items, including ocular and facial involvement, swallowing, speech, limb strength, and forced vital capacity. The total QMG score was obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3) and the score ranges from 0 to 39, with lower scores indicating lower disease activity. A positive change in the score indicates worsening and a negative change indicates improvement.
Time Frame: Baseline and Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 66 | 67
units on a scale | -1.915 (0.682) | -5.398 (0.679) | -6.672 (0.692)
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab ~7 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -3.483, 95% CI 2-sided [-5.614 to -1.584] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Rozanolixizumab ~10 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -4.756, 95% CI 2-sided [-6.821 to -2.859] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline to Day 43 in the Myasthenia Gravis (MG) Symptoms Patient Reported Outcome (PRO) 'Muscle Weakness Fatigability' Score
Description: MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular muscle weakness (items 1-5); bulbar muscle weakness (items 6-15); respiratory muscle weakness (items 16-18); physical fatigue (items 19-33) and muscle weakness fatigability (items 34-42). Study participants were asked to choose response option that how frequently they experienced muscle weakness fatigability (items 34-42) over the past 7 days using a 5-point Likert scale (1="none of the time" to 5="all of the time") for each item. Sum of each item score is linearly transformed to have all domain scores ranging from 0 to 100. Total score is calculated as: (sum of item scores within the scale)/(raw score range) x (total number of items in the scale)/(number of non-missing items in the scale) x100 and ranged from 0 to 100, where higher scores indicated severe symptoms.
Time Frame: Baseline and Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 66 | 67
units on a scale | -10.588 (3.034) | -23.029 (3.034) | -25.751 (3.095)
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab ~7 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -12.441, 95% CI 2-sided [-21.804 to -4.089] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Rozanolixizumab ~10 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -15.163, 95% CI 2-sided [-23.596 to -6.450] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Change From Baseline to Day 43 in the Myasthenia Gravis (MG) Symptoms Patient Reported Outcome (PRO) 'Physical Fatigue' Score
Description: The MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular muscle weakness (items 1-5); bulbar muscle weakness (items 6-15); respiratory muscle weakness (items 16-18); physical fatigue (items 19-33) and muscle weakness fatigability (items 34-42). Study participants were asked to choose the response option that how frequently they experienced physical fatigue (items 19-33) over the past 7 days using a 5-point Likert scale (1="none of the time" to 5="all of the time") for each item. Sum of each item score is linearly transformed to have all domain scores ranging from 0 to 100. Total score is calculated as: (sum of item scores within the scale)/(raw score range) x (total number of items in the scale)/(number of non-missing items in the scale) x100 and ranged from 0 to 100, where higher scores indicated severe symptoms.
Time Frame: Baseline and Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 66 | 67
units on a scale | -10.637 (3.051) | -19.287 (3.046) | -25.459 (3.107)
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab ~7 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.012, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -8.650, 95% CI 2-sided [-18.058 to -0.134] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Rozanolixizumab ~10 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -14.822, 95% CI 2-sided [-23.759 to -5.936] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline to Day 43 in the Myasthenia Gravis (MG) Symptoms Patient Reported Outcome (PRO) 'Bulbar Symptoms' Score
Description: The MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular muscle weakness (items 1-5); bulbar muscle weakness (items 6-15); respiratory muscle weakness (items 16-18); physical fatigue (items 19-33) and muscle weakness fatigability (items 34-42). Study participants were asked to choose response option that best described severity of bulbar muscle weakness (items 6-15) symptoms over past 7 days using a 4-point Likert scale (1="none" to 4="severe") for each item. Sum of each item score is linearly transformed to have all domain scores ranging from 0 to 100. Total score is calculated as: (sum of item scores within the scale)/(raw score range) x (total number of items in the scale)/(number of non-missing items in the scale) x100 and ranged from 0 to 100, where higher scores indicated severe symptoms.
Time Frame: Baseline and Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 66 | 67
units on a scale | -3.519 (2.397) | -14.839 (2.406) | -14.224 (2.464)
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab ~7 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -11.320, 95% CI 2-sided [-18.958 to -4.998] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Rozanolixizumab ~10 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Lehmacher and Wassmer method — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -10.705, 95% CI 2-sided [-17.787 to -3.998] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an AE starting on or after the time of first administration of investigational medicinal product (IMP) up to and including 8 weeks after the last dose.
Time Frame: From Baseline until End of Study Visit (up to Week 14)
Population: The Safety Set consisted of all randomized study participants who received at least one dose of IMP and were analyzed according to the actual treatment the participants received. Two participants randomized to RLZ ~7mg/kg, were administered RLZ ~10mg/kg at baseline visit. So, these two participants were included in RLZ ~7 mg/kg group in randomized set, but in RLZ ~10 mg/kg group in safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 64 | 69
Participants | 45 | 52 | 57

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal of Investigational Medicinal Product (IMP)
Description: A TEAE is defined as an AE starting on or after the time of first administration of IMP up to and including 8 weeks after the last dose.
Time Frame: From Baseline until End of Study Visit (up to Week 14)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 67 | 64 | 69
Participants | 2 | 2 | 4

ADVERSE EVENTS:
Time Frame: From Baseline until End of Study Visit (up to Week 14)
Description: Safety Set was analyzed for TEAEs. Two participants randomized to RLZ ~7mg/kg, were administered RLZ ~10mg/kg at baseline visit. So, these two participants were included in RLZ ~7 mg/kg group in randomized set, but in RLZ ~10 mg/kg group in safety set.
Arm/Group | Placebo | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/64 | 0/69
Serious Adverse Events (participants affected / at risk) | 6/67 | 5/64 | 7/69
Other Adverse Events (participants affected / at risk) | 26/67 | 40/64 | 42/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=67) | Rozanolixizumab ~7 mg/kg (N=64) | Rozanolixizumab ~10 mg/kg (N=69)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Myasthenia gravis crisis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=67) | Rozanolixizumab ~7 mg/kg (N=64) | Rozanolixizumab ~10 mg/kg (N=69)
Diarrhoea (Gastrointestinal disorders) | 9 (14) | 16 (18) | 11 (18)
Nausea (Gastrointestinal disorders) | 5 (12) | 5 (7) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (4) | 1 (3) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 8 (10) | 14 (25)
Nasopharyngitis (Infections and infestations) | 3 (4) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (9) | 4 (4)
Headache (Nervous system disorders) | 13 (31) | 29 (54) | 26 (51)
Hypertension (Vascular disorders) | 0 (0) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03971422/Prot_001.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03971422/SAP_002.pdf